CLINICAL TRIAL: NCT04355273
Title: Effects of Different Concentrations of Pressurized-heparin Flushing Fluid on Coagulation and Platelet Function Monitored by the Sonoclot Analyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20200420
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Heparin; Perioperative
MeSH Terms: interventions — Heparin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heparin with a concentration of 2 U/ml (Experimental): heparin dilution is placed in a pressure bag with a pressure of 300 mmHg
  Interventions: Drug: Heparin
- Heparin with a concentration of 4 U/ml (Experimental): heparin dilution is placed in a pressure bag with a pressure of 300 mmHg
  Interventions: Drug: Heparin
- normal saline (Placebo Comparator): normal saline is placed in a pressure bag with a pressure of 300 mmHg
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Heparin — heparin with a concentration of 2 U/ml is used for pressurized continuous flushing of the invasive arterial pressure monitoring tube
  Arms: Heparin with a concentration of 2 U/ml
Drug: Heparin — heparin with a concentration of 4 U/ml is used for pressurized continuous flushing of the invasive arterial pressure monitoring tube
  Arms: Heparin with a concentration of 4 U/ml
Drug: normal saline — normal saline is used for pressurized continuous flushing of the invasive arterial pressure monitoring tube
  Arms: normal saline

SUMMARY:
Heparin diluent or normal saline is generally used as the arterial tube flushing in clinical practice, but there is no consensus on the choice of flushing fluid. Heparin can affect the blood coagulation function, and even lead to heparin-related thrombocytopenia, increasing the risk of perioperative embolism. Sonoclot is a blood viscoelasticity test, which can provide comprehensive information on the coagulation's cascade and the entire process and be quicker and more effective than routine laboratory coagulation tests. In this research, the coagulation and platelet function analyzer called Sonoclot is used to evaluate the effect of different concentrations of pressurized heparin on the coagulation and platelet function of perioperative patients, which can provide a reference for the clinical choice of appropriate arterial flushing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gastrointestinal cancer
* Ages ranged from 18 to 75
* ASA I~III

Exclusion Criteria:

* Pregnancy
* modified Allen Test negative
* history of taking anti-platelet drugs such as aspirin one week before surgery, heparin allergy and thrombotherapy
* two failed catheterizations of the same artery
* significant diseases in liver and kidney function
* refusal of patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The level of glass bead Activated Clotting Time | through study completion, an average of 3 minute
  10 min after the vein puncture, 2 h after skin incision and at the end of surgery

SECONDARY OUTCOMES:
The level of glass bead Clot Rate | through study completion, an average of 3 minute
  10 min after the vein puncture, 2 h after skin incision and at the end of surgery
The level of glass bead Platelet Function | through study completion, an average of 3 minute
  10 min after the vein puncture, 2 h after skin incision and at the end of surgery
The level of platelet count | through study completion, an average of 2 minute
  24 h after surgery and 48 h after surgery
The frequencies of hand positional changes and manual artery flushing | intraoperative
The amount of infusion volume, blood loss, urine volume | intraoperative
The appearance of local complications of arterial puncture | within 24 h after surgery
  Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China